CLINICAL TRIAL: NCT02267031
Title: The Role of Perioperative Ventilation (Gas Exchange) During Intrabdominal Surgery on Cognitive Function: a Randomized Clinical Study
Brief Title: The Role of Perioperative Ventilation (Gas Exchange) During Intrabdominal Surgery on Cognitive Function
Acronym: ACDYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AC-2012
Record Dates: First submitted 2014-10-02; First posted 2014-10-17 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Response to Hyperoxia; Hypocapnia
Keywords: cognitive dysfunction; mechanical ventilation; hyperoxia; hypocapnia
MeSH Terms: conditions — Hypocapnia; Cognitive Dysfunction; Hyperoxia | interventions — Respiration, Artificial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- normoxia and normocapnia (Active Comparator): Normoxia PaO2 of 70-140 mm Hg Normocapnia PaCO2 of 35-48 mmHg
  Interventions: Procedure: mechanical ventilation
- hyperoxia and normocapnia (Active Comparator): Hyperoxia 150-300 mm Hg Normocapnia PaCO2 of 35-48 mmHg
  Interventions: Procedure: mechanical ventilation
- normoxia and hypocapnia (Active Comparator): Normoxia PaO2 of 70-140 mm Hg Hypocapnia PaCO2 of 25-35 mmHg
  Interventions: Procedure: mechanical ventilation
- hyperoxia-hypocapnia (Active Comparator): Hyperoxia 150-300 mm Hg Hypocapnia PaCO2 of 25-35 mmHg
  Interventions: Procedure: mechanical ventilation

INTERVENTIONS:
Procedure: mechanical ventilation — Patients subjected to scheduled laparoscopic cholecystectomy were enrolled to the ongoing prospective study and randomized into four groups: 1) normoxia and normocapnia (nO2-nCO2), 2) hyperoxia and normocapnia (hO2-nCO2), 3) normoxia and hypocapnia (nO2-lCO2), and 4) hyperoxia-hypocapnia (hO2-lCO2).
  Normoxia PaO2 was referred to PaO2 of 70-140 mm Hg, hyperoxia 150-300 mm Hg, normocapnia PaCO2 of 35-48 mmHg and hypocapnia PaCO2 of 25-35 mmHg.

SUMMARY:
Abdominal surgery commonly requires perioperative relaxation and therefore controlled mechanical ventilation. However, respiratory support can be associated with minor, yet clinically significant changes in blood gas content. The inadvertent hyperoxia (excessively high oxygen) and/or hypocapnia (excessively low carbon dioxide) can result in transient changes in cerebral blood flow and cognitive impair.

DETAILED DESCRIPTION:
The moderate hyperventilation resulting in hypocapnia as well as hyperoxia are common features of mechanical ventilation during general anesthesia. While mild hyperventilation is routinely advocated in laparoscopic surgical interventions, increased FiO2 is set to reinforce safety of respiratory support. Hypocapnia may cause disturbances of cerebral blood flow due to narrowing of cerebral vessels and a decrease cerebral blood flow. Hypocapnia is particularly injurious to the brain in premature infants. Factors that may predispose the immature brain to such injury include poorly developed vascular supply to vulnerable areas, antioxidant depletion by excitatory amino acids, and the lipopolysaccharide and cytokine effects that potentiate destruction of white matter. Data from neonates clearly suggest that severe hypocapnia after hyperventilation contribute to adverse neurologic outcomes. The use of high concentrations of oxygen can lead to a number of events such as the formation of harmful free radicals and activation of lipid peroxidation, resulting in secondary brain injury due to hyperoxia, particularly after suffering anoxia of the brain in resuscitated victims of sudden cardiac arrest. It is recommended to use the fraction of oxygen to maintain saturation at the level of 94-98% when performing cardiopulmonary resuscitation (CPR), due to the risk of reperfusion injury. These disturbances of gas exchange, yet transient can interfere in cerebral blood flow and therefore mental functions.

The primary aim of this study was the assessment of the impact of intraoperative gas exchange (hypocapnia, hyperoxia and their combinations) on the state of higher nervous activity

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age > 18 years and below 80 yrs
* Elective abdominal endoscopic intervention

Exclusion Criteria:

* Known cerebral disorder, incl. traumatic injury and severe vascular impairment
* Known psychiatric illness
* Severe drug or alcohol abuse
* Resent stroke (during last 6 months)
* Pregnancy
* Within the 30 days prior to this study, either entry into any other randomized therapeutic study of an agent not licensed for the intended use or administration of any other investigational agent for the treatment of ALI. Patients must not participate in such studies for at least 30 days after enrolment into this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2012-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 36 hrs
  Cognitive function will be assessed using Montreal Cognitive Assessment Score (MoCA)

SECONDARY OUTCOMES:
Psychological Changes | 6 months
  Using developed phone query (memory, cognition, anxiety etc.)
Pain perception | 6 hrs
  Using Visual Analog Score (VAS)
Pain perception | 36 hrs
  Using Visual Analog Score (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Y. Kirov, MD, PhD, Principal Investigator — Northern State Medical University
Locations (1):
- City hospital # 1 / Northern State Medical University,, Arkhangelsk, Russia